CLINICAL TRIAL: NCT03214055
Title: Effect of Mannitol on Optic Nerve Sheath Diameter in Patients Undergoing Robot-assisted Laparoscopic Radical Prostatectomy: a Prospective Observational Study
Brief Title: Effect of Mannitol on Optic Nerve Sheath Diameter in Patients Undergoing Robotic Prostatectomy
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Kug Kim, Professor, Asan Medical Center
Other Study IDs: 2017-0789
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Mannitol; Diuretics, Osmotic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Mannitol — The mannitol has been administered routinely to prevent renal dysfunction in patients undergoing robot-assisted laparoscopic radical prostatectomy. Participants will receive the mannitol as part of routine medical care, and we will evaluate the change in optic nerve sheath diameters before and after mannitol administration.
  Other Names: Osmotic diuretic

SUMMARY:
We aim to evaluate the change in optic nerve sheath diameters as a surrogate of intracranial pressure before and after mannitol administration in patients who undergo robot assisted laparoscopic radical prostatectomy with pneumoperitoneum and Trendelenburg position.

DETAILED DESCRIPTION:
Mannitol has been frequently used for renal protection during surgery. Optic nerve sheath diameter is used to evaluate intracranial pressure noninvasively. Robot-assisted laparoscopic radical prostatectomy can induce an increase in optic nerve sheath diameter due to Trendelenburg position and carbon dioxide insufflation. We therefore aim to evaluate the change in optic nerve sheath diameters before and after mannitol administration in patients who undergo robot assisted laparoscopic radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* prostate cancer patients undergoing robot assisted laparoscopic radical prostatectomy.
* 20 year old or above, 79 year old or below.
* agreed to participate this study.

Exclusion Criteria:

* history of cerebrovascular accident.
* history of congestive heart failure.
* history of pulmonary edema.
* history of anaphylaxis to mannitol.
* conversion to open prostatectomy.
* combined with other operation.
* inability to measure optic nerve sheath diameter.

Ages: 20 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male included.
Study Population: Prostate cancer patients who undergo Robot-assisted laparoscopic radical prostatectomy.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-20 (Actual)

PRIMARY OUTCOMES:
Change in optic nerve sheath diameters | 5 minutes after pneumoperitoneum and Trendelenburg position, 90 minutes after mannitol administration during pneumoperitoneum and Trendelenburg position
  Change in optic nerve sheath diameters before and after mannitol administration

SECONDARY OUTCOMES:
Change in optic nerve sheath diameters | 5 minutes after pneumoperitoneum and Trendelenburg position, 60 minutes after mannitol administration during pneumoperitoneum and Trendelenburg position
  Change in optic nerve sheath diameters before and after mannitol administration
Change in optic nerve sheath diameters | 5 minutes after pneumoperitoneum and Trendelenburg position, 30 minutes after mannitol administration during pneumoperitoneum and Trendelenburg position
  Change in optic nerve sheath diameters before and after mannitol administration
Optic nerve sheath diameter | 10 minutes after induction of anesthesia
  Optic nerve sheath diameter before mannitol administration
Optic nerve sheath diameter | Intraoperative (during skin closure)
  Optic nerve sheath diameter after mannitol administration

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kug Kim, MD,PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No